CLINICAL TRIAL: NCT00636740
Title: A Multi-Center Phase II Study to Compare MER-101 (20mg) Tablets To Intravenous Zometa 4mg in Male Bisphosphonate-Naive Hormone Refractory Prostate Cancer Patients
Brief Title: Multi-Center Phase II Study to Compare MER-101 20mg Tablets to Intravenous Zometa 4mg in Male Bisphosphonate-Naive, Hormone Refractory Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merrion Pharmaceuticals, LLC (Industry)
Responsible Party: Thomas W. Leonard, PhD, Merrion Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MER-101-03
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Hormone-Refractory Prostate Cancer
Keywords: Prostate cancer, hormone resistant, bisphosphonate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Experimental): MER-101 20mg Tablets Regimen 1
  Interventions: Drug: Zoledronic Acid 20mg Tablets
- C (Experimental): MER-101 20mg Tablets Regimen 2
  Interventions: Drug: Zoledronic Acid 20mg Tablets
- A (Active Comparator): Zometa Injection
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid 20mg Tablets — Oral enteric coated tablets, 20mg, weekly, 8 weeks
  Other Names: MER-101
  Arms: B
Drug: Zoledronic Acid — Zoledronic Acid infusion, 4mg, every 4 weeks for 8 weeks
  Other Names: Zometa
  Arms: A
Drug: Zoledronic Acid 20mg Tablets — Oral enteric coated tablets, 20mg, once a day for 4 consecutive days during week 1, weekly for weeks 5, 6, 7, 8
  Other Names: MER-101
  Arms: C

SUMMARY:
The objective of MER-101-03 is to examine the effects of two different dosing regimens of MER-101 20mg tablets versus Zometa 4mg IV infusion once-monthly therapy. The effects will be monitored on a weekly basis by measuring various markers of bone metabolism. Patients to be enrolled will be those who have not received any previous bisphosphonate therapy. The study will be carried out on prostate cancer patients who are no longer on hormone therapy. Treatment in the study will be for a 2-month period.

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer with rising PSA levels after hormone treatment and bone metastasis based on an X-ray.

Exclusion Criteria:

* Already be on a bisphosphonate treatment (Zometa, Fosamax, Actonel)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Effects on 4 markers of bone metabolism | Weekly

SECONDARY OUTCOMES:
Brief Pain Inventory | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Leonard, PhD, Study Director — Merrion Pharmaceuticals, LLC
Locations (13):
- United States (8):
  - Birmingham Hematology & Oncology Associates, LLC, Birmingham, Alabama
  - Cancer Care of North Florida, P.A., Lake City, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Green Clinic, LLC, Ruston, Louisiana
  - New York Urological Associates, PC, New York, New York
  - Charleston Hematology Oncology Associates, PA, Charleston, South Carolina
  - Cancer Outreach Associates, P.C., Abingdon, Virginia
- Estonia (3):
  - East Tallinn Central Hospital, Tallinn
  - North Estonian Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Latvia (2):
  - O. Hublarovs Private Practice, Daugavpils
  - P. Stradina Clinical University Hospital, Riga